CLINICAL TRIAL: NCT06089447
Title: A Pilot Randomised Controlled Trial of 'The Shadow of Tallystick Valley' for Children and Young People Experiencing Family Substance Use
Brief Title: A Pilot Randomised Controlled Trial of Intervention for Children and Young People Experiencing Family Substance Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Surrey (Other)
Responsible Party: Principal Investigator, India Smith, Trainee Clinical Psychologist, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FHMS 22-23 237 EGA
Record Dates: First submitted 2023-10-03; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Wellness, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Masking Description: The children and young people will not know which group they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Participants will receive the intervention immediately
  Interventions: Behavioral: A story based intervention called 'The Shadow of Tallystick Valley'
- Waitlist Group (Active Comparator): Participants will be allocated to a waitlist group and will receive the intervention aft 6 months.
  Interventions: Behavioral: A story based intervention called 'The Shadow of Tallystick Valley'

INTERVENTIONS:
Behavioral: A story based intervention called 'The Shadow of Tallystick Valley' — 'The Shadows of Tallystick Valley' is a story based intervention for CYP aged 7 - 14 years aimed at supporting the psychological wellbeing and resilience of those affected by familial substance misuse. It has been designed by Book of Beasties, a developer of games and educational content, in collaboration with the charity Change Grow Live, who support those experiencing substance misuse and CYP affected by familial substance misuse in the UK. The wellbeing resource harnesses protective factors, such as respectful and caring conversations with professionals (Wangansteen and Westby, 2019), to facilitate a safe and supportive environment aimed towards understanding the CYPs experience, support their psychological wellbeing and building resilience and coping skills. It uses fictional narratives, including characters that represent particular topics which act as drivers for engagement.

SUMMARY:
The study is investigating the feasibility and acceptability of the story-based intervention, The Shadows of Tallystick Valley, aimed at improving the psychological wellbeing and resilience of children and young people who are affected by familial substance use. A secondary aim of the study is to identify whether there is a 'signal of efficacy'. The early intervention is a story and activity book designed and developed by Book of Beasties, in collaboration with the charity Change Grow Live (CGL), who work directly with children and young people experiencing familial substance use. The intervention is used by s at CGL with children and young people engaged with the service. In the present study, we aim to evaluate the story-based intervention within a pilot randomised controlled trial. Participants will be randomised to either receive the intervention or to join a waitlist for the same intervention. The effects of the story-based intervention will be assessed using pre and post psychological well-being and resilience measures, including KidCOPE, the Stirling Children's Wellbeing Scale and the Child and Youth Resilience Measure. The primary outcome measures are concerned with overall psychological wellbeing.

DETAILED DESCRIPTION:
The aims of this pilot trial are as follows:

To determine whether a full trial is justified; To determine the feasibility and acceptability of the story-based intervention in improving psychological wellbeing and emotional literacy in children and young people experiencing familial substance use; To establish the effect size on the co-primary outcomes for a sample size calculation for a definitive trial.

To establish the feasibility of the intervention, we will collect data on the primary outcome for at least 80% of the recruitment target, and have an attrition rate that does not exceed 40%. A definitive trial will be justified if we are able to successfully recruit and retain participants in the trial, and if both the trial procedures and intervention are deemed to be acceptable to participants. Although the primary aim of pilot RCTs is to answer questions related to feasibility, an important secondary aim is to determine whether there is a signal of efficacy so as to inform the decision to progress to a definitive trial (Beets et al., 2021). The between-group effects will determine whether there is a signal of efficacy in favour of the Shadow of Tallystick Valley intervention and further support the need for a definitive randomised controlled trial (RCT). A signal of efficacy will be considered to be found if the between-group effect size on the co-primary outcomes is in favour of the intervention. Where these conditions are met, this study will therein provide the parameters needed to estimate the sample size for a definitive RCT. We will assess whether the study design is acceptable to participants using recruitment and retention rates (i.e., study and intervention uptake and dropout rates) and qualitative interviews with participants.

The intervention will be offered to children and young people already connected with CGL. Children and young people are referred to the service via a referral from an adult known to them. This can include (but is not limited to) family members, social workers, teachers, school staff, substances, or other youth worker professionals.

Recruitment methods:

Study advert and information pack will be shared by staff across the service with all children and young people who meet the inclusion criteria. If the child or young person wants to proceed, both they and their parent or caregiver must provide either written or verbal consent. Consent will be collected by the assigned support worker at Change Grow Live.

If in the instance a participant withdraws their consent, they will have two weeks after the intervention has been delivered to do so and relevant data will be removed and destroyed. Beyond the two week mark, the data will be written up. If a parent/ caregiver withdraws their consent, CGL would discuss the parents' concerns with them in the hope they can resolve them. If parents/caregiver consent is still withdrawn and the child is under 13, the participant will no longer be involved in the study and relevant data will be destroyed. If in the instance the parent/caregiver withdraws consent for a young person who is over 13 years of age and Gillick Competent, the young person will be able to continue in the study. This is inline with CGL's policy and procedures. If in the instance the parent / caregiver withdraws consent for a child below the age of 13 years, the child or young person will be withdrawn from the study.

The target sample size is based on guidelines by Whitehead et al. (2015) for a pilot trial prior to a main trial with 90% power and two-sided 5% significance expecting a small to medium effect size. We plan to recruit 25 participants per arm (50 in total).

Experimental Design

The present study is a single-blind external pilot randomised controlled trial with two parallel arms including optional qualitative feedback. Support Workers will children and young people (aged between 7 and 18 years). Interested participants will be given a participant information sheet. After reading the PIS, if potential participants are interested in participating in the trial, they will complete an eligibility assessment to determine whether they meet the inclusion/exclusion criteria. If the participant meets the eligibility criteria, they will be invited to complete a consent form. Prospective participants will not be able to progress in the trial without completing the consent statement.

Once participants have provided consent and consent has been given from parent/carer, participants will be allocated a unique ID code and asked to complete the baseline (T0) assessment. A file linking the participants' contact information with the unique IDs will be stored securely in a password-protected file in a OneDrive folder held on the University of Surrey's system. The PI will have the password for this file and give access to this to other members of the research team as needed. The password will not be shared outside of the research team. The T0 assessment can be completed either online or in person. There will be video instructions on how to complete the questionnaires for children and young people to then complete them independently. These videos will be produced after ethical approval so that the information conveyed is in line with the approved protocol and study materials. After the T0 assessment has been completed, participants will be randomly allocated to either receive the immediate intervention arm or a wait-list control group. The outcome of this randomisation will be emailed to the PI and will be logged in the secure, password protected file. The randomisation will be conducted using the simple randomisation function available from Sealed Envelope. Participants will not know which arm they have been allocated to. The support workers will deliver the intervention with the children and young people allocated to the control group of the study. They will have received at least one full day of training designed and delivered by CGL's National Hidden Head Lead. Participants will be contacted 18 weeks post-randomisation to complete the T1 assessment. The T1 assessment can be completed in person or online depending on participants preference. The T1 assessment will replicate the T0 assessment. After completing the T1 assessment, participants will be presented with an end of trial debrief statement.

Data Collection The trial will utilise a mixed methods approach, collecting both quantitative and qualitative data. The quantitative data will be collected at T0 and T1. The qualitative data will be collected from the intervention group in the form of written feedback form or an audio recording after the T1 assessment. Data collection should not involve contact with adults outside of CGL but must have independence to allow for adequate blinding. The data can be collected either online via Qualtrics or in hard copy. There is the potential to have video instructions on how to complete the questionnaires for children and young people to then complete them independently.

The main trial data will be entered into SPSS by the principal investigator. The items will be coded and scored in line with the original questionnaire protocols. A random selection of 20% of the data will be checked against the source (i.e. hard copies of questionnaires) to ensure data quality.

The Principal Investigator will act as the data custodian. The data will be owned by the lead organisation, the University of Surrey.

Data analysis All of the variables will be summarised using descriptive statistics by arm at each time point. We will calculate Cohen's d between-group effect sizes with 95% confidence intervals, comparing the T1 scores of the intervention versus control arms, adjusting effects for the baseline scores using an ANCOVA. The level of missing data for all outcome measures will be reported. As the present study is a pilot trial, we will not be testing any hypotheses and are instead testing evidence for a signal of efficacy in the desired direction.

The research process data will be used to understand the rates of recruitment and retention at all stages of the study. We will report the number of participants who completed and dropped out at each stage of the trial in the form of a CONSORT diagram. The quantitative adherence data will be the number of sessions completed with a child or young person and used to understand the degree of engagement with the intervention amongst participants. We will report the responses using descriptive statistics and describe any patterns that can be observed.

All of the data collected over the course of the study will be collected, stored and maintained in line with the General Data Protection Regulation (GDPR) (Information Commissioner's Office, 2018) . Any hard copies will be scanned so as to become electronic documents. The hard copies will be destroyed. Electronic documents/data will all be stored within a University of Surrey OneDrive folder and protected with a password, accessed only by the research team. The PI will have all of the passwords and share these with members of the research team as needed. No one outside of the research team will have access to the passwords. The PI will assume responsibility for ensuring adherence to the data security protocol.

Data will be retained in accordance with the General Data Protection Regulation (GDPR) (Information Commissioner's Office, 2018) and (Medical Research Council, 2012) policies on data storage and archiving. Once the data analysis has been finalised, all anonymised data will be archived at the University of Surrey for up to 10 years. The anonymised data will be retained indefinitely by the PI.

Ethical considerations Consent to take part in this study will be informed. All participants and parents/carers of participants will be given the Participant Information Sheet (PIS) and will not be limited in terms of the amount of time they want to read through it. All participants will be told within the PIS and the consent forms that they can withdraw from the research study at any point. Participants will be asked to sign an item on the consent form that confirms that they are aware of their right to withdraw, and that they are not obligated to provide a reason for leaving the study.

All of the data collected within the research study will be treated as confidential. Identifiable data will not be shared outside of the research team. The study will comply with the General Data Protection Regulation (GDPR) and Data Protection Act 2018, which require data to be de-identified as soon as it is practical to do so. Participants will be identified on all documents (both hard copy and electronic) containing research data using a unique participant ID code. All documents will be stored securely and only accessible by the research team. The research team will safeguard the privacy of participants' data.

Participants will be informed within the PIS and consent form that anything they share over the course of the study will be treated as confidential, except for where this information puts themselves or other people at risk. Where confidentiality needs to be broken for safeguarding reasons, the information will only be shared with persons who have a responsibility to monitor and minimise this risk (e.g. s, personal tutors, university counselling team, local safeguarding authorities, mental health services). Participants will be asked to sign an item on the consent form that confirms that they understand our confidentiality policy.

Participants will be reimbursed for their time and effort at a rate of £5 for pre and £5 for post questionnaires completed (£10 in total) in the form of vouchers.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7 - 14 years;
* Child: 7 - 10
* YP: 11 - 14
* Able to read age appropriate materials independently;
* Have someone in their family using alcohol and/or substances;
* Have received parental/caregiver consent to take part in the study;
* Have an assigned support worker

Exclusion Criteria:

* They are below age 7 years or above 14 years;
* They are currently engaging in self-harm, including all forms of self harm as set out by Mind (2020), and/or have plans to end their life;all forms of self harm
* Have not given consent to take part in the study;
* Have not received parent or caregiver consent to take part in the study.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Stirling Children's Wellbeing Scale (SCWBS) | Two weeks
  The Stirling Children's Wellbeing Scale (SCWBS) (Liddle and Carter, 2015) is a 15-item questionnaire measuring wellbeing.

SECONDARY OUTCOMES:
KidCOPE | Two weeks
  Kidcope (Spirito et al., 1988) is a brief, clinical checklist designed to screen cognitive and behavioural coping in children and adolescents. The checklist covers problem-solving, distraction, social support, social withdrawal, cognitive restructuring, self-criticism, blaming others, emotional expression, wishful thinking, and resignation.
Child and Youth Resilience Measure | Two weeks
  The Child & Youth Resilience Measure (Ungar and Liebenberg, 2011) is a 12 item questionnaire that measures overall resilience, as well as three subcategories that influence resilience processes; individual traits, relationship to caregiver(s), and contextual factors that facilitate a sense of belonging

CONTACTS AND LOCATIONS:
Overall Officials: India Smith, Principal Investigator — Student
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data may be shared outside of the research team for research purposes. Participants will be asked to provide written consent (either electronically or in hard copy) for their anonymous data to be shared in this way. Where an academic journal requires that the original data is made available as per their publication terms, the research team will share only the anonymised data set - this type of data sharing will be covered under the consent form item related to 'data sharing for research purposes'. Data will not be shared with the parent or caregiver.
  Any requests to access the anonymised trial data should be made to the PI. Data must not be shared outside the research team without the permission of the PI. All members of the research team have been made aware of and have agreed to abide by this data sharing policy. The PI reserves the right to reject any requests to access the anonymised trial data.

REFERENCES:
- [Background] Beets MW, von Klinggraeff L, Weaver RG, Armstrong B, Burkart S. Small studies, big decisions: the role of pilot/feasibility studies in incremental science and premature scale-up of behavioral interventions. Pilot Feasibility Stud. 2021 Sep 10;7(1):173. doi: 10.1186/s40814-021-00909-w. PMID 34507624
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Information Commissioner's Office. (2018). Guide to the General Data Protection Regulation (GDPR). https://ico.org.uk/for-organisations/guide-to-the-general-data-protection-regulation-gdpr
- [Background] Medical Research Council. (2012). Good research practice: Principles and guidelines. In MRC ethics series.
- [Background] Mind. (2020). Self Harm. Accessible via self-harm-2020.pdf (mind.org.uk)